CLINICAL TRIAL: NCT01369121
Title: A Phase I/II Open Label Individual Dose Titration Trial of the Human Corticotropin- Releasing Factor (hCRF), Corticorelin Acetate Injection (Xerecept®), to Determine the Tolerability of Xerecept® in a Pediatric Population
Brief Title: Tolerability Study of Xerecept® in Pediatric Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Single subject remained on study - transferred to compassionate use
Sponsor: Celtic Pharma Development Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDS 1001
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Brain Edema; Brain Tumor
Keywords: peritumoral brain edema; edema; malignant brain tumor; brain tumor; dexamethasone; Decadron
MeSH Terms: conditions — Brain Edema; Brain Neoplasms; Edema | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xerecept (Experimental): All patients will receive hCRF (XERECEPT)
  Interventions: Drug: XERECEPT

INTERVENTIONS:
Drug: XERECEPT — BID dosing, subcutaneous for 1 year
  Other Names: hCRF; Corticorelin acetate injection

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of Xerecept® in children with central nervous system tumors and to identify appropriate doses of Xerecept® to be used in subsequent pediatric clinical trials.

DETAILED DESCRIPTION:
Steroid-related side effects are much more severe in a pediatric population than they are in adults. The side effects appear more quickly and are often apparent in as few as 14 days. Dexamethasone side effects in children include rounding of the face, acne, increased body hair, muscle weakness, osteoporosis, mood changes, weight gain, fluid retention, glucose instability, high blood pressure, increased susceptibility to infection, stunted growth and aseptic necrosis of the hip joints14-16.

Although extensive studies have been performed with Xerecept® in adults, no studies have been performed with Xerecept® in pediatric subjects. Therefore, this study is being conducted to evaluate the safety and tolerability of Xerecept® in children with central nervous system tumors and to identify appropriate doses of Xerecept® to be used in subsequent pediatric clinical trials. The study will also explore if Xerecept®, when administered to pediatric patients, is effective in allowing decreases in dexamethasone dosing

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed primary, recurrent or metastatic cerebral tumors and require chronic steroid dosing to manage symptoms of peritumoral brain edema (No histological confirmation is required of optic pathway tumors or brain stem gliomas)
2. Have been taking dexamethasone (or equivalent) at a dose of ≥1 mg/day for a minimum of 14 days and have had a stable dose for at least 7 days.
3. Have one or more steroid-associated side effects at Screening (See Appendix A1 for a list of qualifying events)
4. Capable of self-administration of subcutaneous injections twice daily or availability of assistance from caregiver.
5. Karnofsky/Lansky performance status ≥ 40
6. Life expectancy of at least 6 months
7. Female subjects must not be pregnant or breast-feeding and, if of childbearing potential, must use adequate methods of contraception during the study

10. Ability to provide written informed consent or, if unable to provide, have a legal guardian or representative provide written informed

Exclusion Criteria:

1. Evidence of previous or current overt renal, hepatic or pulmonary diseases or active uncontrolled infection
2. Subject and/or parent/guardian is unwilling or unable to comply with this protocol
3. Subject has a known history of allergy or intolerance to hCRF or other ingredients in the Xerecept® solution (e.g., methionine, mannitol)
4. Subject has a known history of hepatitis C virus, hepatitis B surface, or human immunodeficiency virus (HIV).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 months
  To define the maximum tolerated dose (MTD) of Xerecept® in pediatric patients; the MTD will be defined as the dose at which 1 or fewer of six patients experiences a dose limiting adverse event of any kind.

SECONDARY OUTCOMES:
Dexamethasone Dosing | 1 Year
  To explore if Xerecept®, when administered to pediatric patients, is effective in allowing decreases in dexamethasone dosing
Incidence and severity of specified Steroid-Related Side Effects | 1 year
  To explore the clinical benefit associated with a reduction in steroid dosing over the course of the study by comparing the incidence and severity of pre-specified steroid-related side effects in all patients.
Number of patients with adverse events | 1 Year
  Adverse events will be recorded at each study visit and detailed by SOC to define the safety profile of Xerecept in pediatric patients
Change from baseline in clinical chemistry, hematology and urinalysis measures | 1 Year
  Standard clinical chemistry, hematology and urinalysis measures will be analyzed at baseline and monthly during the study; changes from baseline will be measured over the course of the study
PedsQL™ Quality of Life Inventory Scores | 1 Year
  Child self report and parent proxy reports conducted at each study visit to assess changes in health-related quality of life over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Children's Memorial Hospital, Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Dana-Farber Cancer Institute Pediatric Oncology, Boston, Massachusetts